CLINICAL TRIAL: NCT04507776
Title: Long Term Adherence and Efficacy of Etanercept in SpA Iraqi Patients: 7 Year Data From Local Registry
Brief Title: Study To Evaluate The Efficacy And Long-Term Adherence Of Spondyloarthropathies(SpA) Patients On Enbrel
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801414
Record Dates: First submitted 2020-07-27; First posted 2020-08-11 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Spondyloarthrosis
MeSH Terms: conditions — Spondylarthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with spondyloarthropathies: Patients with spondyloarthrosis that received Etanercept as treatment for disease
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Patients with spondyloarthrosis as provided in real world practice
  Other Names: Enbrel

SUMMARY:
This study is to evaluate local data in Iraqi patients with Spondyloarthropathies on Enbrel treatment with regards to efficacy and adherence using data from the Baghdad Teaching Hospital (Rheumatology Center)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed SpA patients
* 18 years of age and older.
* Did not receive previous other biological treatments.
* Patients have at least 1 year on Enbrel.

Exclusion Criteria:

* Had previously used another biological treatments.
* Use of etanercept for less than 1 year duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients data from the local Baghdad Teaching Hospital (Rheumatology Center) registry
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Younis AA, Al-Hafidh AH, Adnan A, Yasiry D, Abdulateef N, Gorial FI, Llamado L, AlJabban A. Long-Term Adherence to Etanercept in Treatment Effectiveness of Patients with Spondyloarthritis: 7-Year Data from the Iraq National Registry. Rheumatol Ther. 2022 Dec;9(6):1605-1616. doi: 10.1007/s40744-022-00497-y. Epub 2022 Sep 30. PMID 36178583
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data of Iraq's participants aged greater than or equal to (>=) 18 years, who received etanercept for at least 1 year, anytime from May 2012 through August 2019, for treatment of spondyloarthropathies (SpA) and met American College of Rheumatology/ European League Against Rheumatism (EULAR) 2019 criteria for SpA were included in the study. Data were collected from dermatology center of Baghdad teaching hospital. Available data were evaluated in 1 month of this retrospective, observational study.
Groups:
- Etanercept: Participants with SpA received etanercept for at least 1 year (anytime from May 2012 to August 2019) under standard real world clinical practice. Data of these participants were studied for 1 month in this retrospective, observational study.
Period: Overall Study
Arm/Group | Etanercept
Started | 763
Completed | 562
Not Completed | 201
Not completed — Participants did not meet the entrance criteria | 201

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants whose data were included in the study for retrospective observation.
Arm/Group | Etanercept
Number analyzed (Participants) | 763
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 627
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 7 Years Adherence to Etanercept
Description: In this outcome measure, percentage of participants who continued etanercept treatment and adhered to the treatment for 7 years were reported.
Time Frame: 7 years [from the data retrieved and observed in 1 month of this study]
Population: Analysis population included all participants whose data were included in the study for retrospective observation.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 763
Percentage of participants | 60.6

2. Other Pre Specified Outcome: Absolute Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Baseline and Last Visit: Participants Adherent and Not Adherent to Treatment
Description: BASDAI is a set of 6 questions to determine disease activity in participant with SpA. Participants answered each 6 questions on a scale of 0 (no problem) to 10 (the worst problem). The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score is then divided by 5. BASDAI score = (Q1 + Q2 + Q3+ Q4+ [Q5 + Q6/2])/5. BASDAI score ranges from 0 (best) to 10 (worst), where higher scores meant worse condition. This outcome measure compared absolute BASDAI score between the participants who were adherent and not adherent to treatment. Comparison was done for 1 and 7 year adherence. For Year 1 adherence, last visit was Year 1 (Month 12). For Year 7 adherence last visit was Year 7.
Time Frame: Year 1 adherence: Baseline (pre-treatment), Year 1; Year 7 adherence: Baseline (pre-treatment), Year 7 [from the data retrieved and observed in 1 month of this study]
Population: Analysis population included all participants whose data were included in the study for retrospective observation. Here, "number analyzed" signifies the number of participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Etanercept: Participants Adherent to Treatment: Participants with SpA received etanercept for at least 1 year (anytime from May 2012 to August 2019) under standard real world clinical practice and were adherent to treatment. Data of these participants were studied for 1 month in this retrospective, observational study.
- Etanercept: Participants Not Adherent to Treatment: Participants with SpA received etanercept for at least 1 year (anytime from May 2012 to August 2019) under standard real world clinical practice and were not adherent to treatment. Data of these participants were studied for 1 month in this retrospective, observational study.
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 700 | 63
Units on a scale
  Year 1 Adherence: Baseline | 8.0579 (0.83161) | 8.0238 (0.81532)
  Year 1 Adherence: Year 1 (Month 12) | 1.3310 (1.74750) | 3.8261 (1.71364)
  Year 7 Adherence: Baseline: number analyzed (Participants) | 80 | 52
  Year 7 Adherence: Baseline | 8.4813 (0.51830) | 8.0000 (0.88561)
  Year 7 Adherence: Year 7: number analyzed (Participants) | 80 | 50
  Year 7 Adherence: Year 7 | 1.3256 (1.49022) | 1.1040 (1.68353)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 1 Adherence: Baseline; Test type: Other; p = 0.75, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 1 Adherence: Year 1 (Month 12); Test type: Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 7 Adherence: Baseline; Test type: Other; p < 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 7 Adherence: Year 7; Test type: Other; p = 0.43, t-test, 2 sided

3. Other Pre Specified Outcome: Change From Baseline in BASDAI Score at Last Visit: Participants Adherent and Not Adherent to Treatment
Description: BASDAI is a set of 6 questions to determine disease activity in participant with SpA. Participants answered each 6 questions on a scale of 0 (no problem) to 10 (the worst problem). The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score is then divided by 5. BASDAI score = (Q1 + Q2 + Q3+ Q4+ [Q5 + Q6/2])/5. BASDAI score ranges from 0 (best) to 10 (worst), where higher scores meant worse condition. This outcome measure compared change from baseline in BASDAI score at last visit between the participants who were adherent and not adherent to treatment. Comparison was done for 1 and 7 year adherence. For Year 1 adherence, last visit was Year 1 (Month 12). For Year 7 adherence last visit was Year 7.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Etanercept: Participants Adherent to Treatment; Etanercept: Participants Not Adherent to Treatment: Participants with SpA received etanercept for at least 1 year (anytime from May 2012 to August 2019) under standard real world clinical practice. Data of these participants were studied for 1 month in this retrospective, observational study.
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 700 | 63
Units on a scale
  Year 1 Adherence: Change at Year 1 (Month 12) | 6.7269 (1.90446) | 4.1977 (1.84639)
  Year 7 Adherence: Change at Year 7: number analyzed (Participants) | 80 | 52
  Year 7 Adherence: Change at Year 7 | 6.8344 (1.86489) | 6.4096 (2.30636)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 1 Adherence: Change at Year 1 (Month 12); Test type: Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 7 Adherence: Change at Year 7; Test type: Other; p = 0.247, t-test, 2 sided

4. Other Pre Specified Outcome: Absolute Bath Ankylosing Spondylitis Functional Index (BASFI) Score at Baseline and Last Visit: Participants Adherent and Not Adherent to Treatment
Description: BASFI is a set of 10 questions to determine degree of functional limitation in participants with SpA. Participants answered each 10 questions on a scale of 0 (no functional impairment) to 10 (maximal impairment). BASFI score was calculated as mean of scores from 10 questions. BASFI score ranged from 0 (no functional impairment) to 10 (maximal impairment), where higher scores meant worse condition. This outcome measure compared absolute BASFI score between the participants who were adherent and not adherent to treatment. Comparison was done for 1 and 7 year adherence. For Year 1 adherence, last visit was Year 1 (Month 12). For Year 7 adherence, last visit was Year 7.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 700 | 63
Units on a scale
  Year 1 Adherence: Baseline | 7.7324 (1.13568) | 7.9143 (0.93668)
  Year 1 Adherence: Year 1 (Month 12) | 1.3028 (1.69316) | 3.7372 (1.71182)
  Year 7 Adherence: Baseline: number analyzed (Participants) | 80 | 52
  Year 7 Adherence: Baseline | 6.6812 (1.60341) | 7.8058 (0.98626)
  Year 7 Adherence: Year 7: number analyzed (Participants) | 80 | 50
  Year 7 Adherence: Year 7 | 1.3256 (1.49022) | 0.9720 (1.39840)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 1 Adherence: Baseline; Test type: Other; p = 0.21, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 1 Adherence: Year 1 (Month 12); Test type: Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 7 Adherence: Baseline; Test type: Other; p = 0.62, t-test, 2 sided
Statistical Analysis 4: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Year 7 Adherence: Year 7; Test type: Other; p = 0.18, t-test, 2 sided

5. Other Pre Specified Outcome: Change From Baseline in BASFI Score at Last Visit: Participants Adherent and Not Adherent to Treatment
Description: BASFI is a set of 10 questions to determine degree of functional limitation in participants with SpA. Participants answered each 10 questions on a scale of 0 (no functional impairment) to 10 (maximal impairment). BASFI score was calculated as mean of scores from 10 questions. BASFI score ranged from 0 (no functional impairment) to 10 (maximal impairment), where higher scores meant worse condition. This outcome measure compared change from baseline in BASFI score at last visit between the participants who were adherent and not adherent to treatment. Comparison was done for 1 and 7 year adherence. For Year 1 adherence, last visit was Year 1 (Month 12). For Year 7 adherence last visit was Year 7.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 700 | 63
Units on a scale
  Year 1 Adherence: Change at Year 1 (Month 12) | 6.4296 (2.03555) | 4.1771 (1.88158)
  Year 7 Adherence: Change at Year 7: number analyzed (Participants) | 80 | 52
  Year 7 Adherence: Change at Year 7 | 5.1206 (2.38577) | 6.3327 (1.94510)
Statistical Analysis 1: Comparison: Etanercept vs Etanercept: Participants Not Adherent to Treatment; Year 1 Adherence: Change at Year 1 (Month 12); Test type: Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Etanercept: Participants Not Adherent to Treatment; Year 7 Adherence: Change at Year 7; Test type: Other; p = 0.003, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events not collected during the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT04507776/Prot_SAP_000.pdf